CLINICAL TRIAL: NCT04423627
Title: Sympathetic Regulation of Large Artery Stiffness in Humans With Age-Related Isolated Systolic Hypertension
Brief Title: Sympathetic Regulation of Large Artery Stiffness in Humans With ISH
Acronym: SELECT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Gary L. Pierce, PhD, Associate Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202004244
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Hypertension, Systolic; Stiffness, Aortic
MeSH Terms: conditions — Isolated Systolic Hypertension | interventions — Clonidine; Hydrochlorothiazide

STUDY DESIGN:
Intervention Model Description: Randomized, placebo controlled, parallel design
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Clonidine (Experimental): 0.2 mg/day oral
  Interventions: Drug: Clonidine
- Hydrochlorothiazide (Active Comparator): 37.5 mg/day oral
  Interventions: Drug: Hydrochlorothiazide
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clonidine — Clonidine 0.2 mg/day oral tablet
  Arms: Clonidine
Drug: Hydrochlorothiazide — Hydrochlorothiazide 37.5 mg/day oral tablet
  Arms: Hydrochlorothiazide
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Stiffening of your blood vessels, particularly the large vessels from your heart (called the aorta and carotids) you age contributes to the development of cardiovascular disease (CVD) such as heart attack and stroke. Nerve activity from your brain to your body also increases with advancing age but it is unknown if this nerve activity contributes directly to the stiffening on your blood vessels in older adults in addition to high blood pressure. Therefore, successful completion of the proposed aims will have a significant clinical impact by identifying if nerve activity from your brain could be a novel target for therapies that would lower stiffness of the aorta and carotid arteries in older adults.

ELIGIBILITY:
Inclusion Criteria:

* age 60-85
* non-smoking
* clinically healthy
* untreated or treated stage 1 isolated systolic hypertension (ISH) (systolic BP 130-139 mmHg; diastolic BP <90 mmHg) or stage 2 ISH (systolic BP 140-159 mmHg; diastolic BP <90 mmHg) per 2017 AHA/ACC hypertension guidelines
* if subject is on antihypertensive medications, they will stop taking medication for a one-week washout period after Visit 1 before they return for Visit 2. They will come in at day 3 and day 7 of the one-week washout for a BP reading, to confirm that systolic BP is <160 mmHg.

Exclusion Criteria:

* no history of cardiovascular disease (e.g., myocardial infarction, bypass surgery, angioplasty/stent, heart failure, cardiomyopathy, pacemaker/defibrillator, peripheral artery disease), pulmonary disease, liver disease, Type I or II diabetes, cancer (treated by chemotherapy and/or radiation), psychiatric illness, on aspirin or other non-steroidal anti-inflammatory drugs (NSAIDs).
* aspirin, NSAIDs, vitamins, herbal supplements, omega-3-fatty acids will have to discontinue for at least 1 week before participation and remain discontinued during the study.
* blood thinners, serotonin reuptake inhibitors (SSRIs), or PDE5 inhibitors will also be excluded.
* Women must be postmenopausal for at least 6 months (surgical or natural) and not currently on hormone replacement therapy.
* Subjects not on antihypertensive will not be eligible if their resting clinic systolic BP is <130 mmHg or >160 mmHg and diastolic BP >90 mmHg.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Change in carotid-femoral pulse wave velocity | Baseline and after 4 weeks
  Aortic stiffness

SECONDARY OUTCOMES:
Change in carotid distensibility index | Baseline and after 4 weeks
  Change in carotid distensibility
Change in carotid flow pulsatility index | Baseline and after 4 weeks
  Change in carotid flow pulsatility
Change in carotid intimal medial thickness (IMT) | Baseline and after 4 weeks
  Change in carotid wall thickness

CONTACTS AND LOCATIONS:
Overall Officials: Gary Pierce, PhD, Principal Investigator — University of Iowa
Locations (2):
- United States (2):
  - Amy Stroud, Iowa City, Iowa
  - University of Iowa, Iowa City, Iowa

IPD SHARING:
Plan to Share IPD: No